CLINICAL TRIAL: NCT01307111
Title: A Randomized Control Trial of Misoprostol Versus Placebo for Cervical Priming in IUD Insertion for Nulliparous Women
Brief Title: Misoprostol Prior to Intrauterine Device (IUD) Insertion in Nulliparous Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Eve Espey, Professor, OB-GYN, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRRC #09-426
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-02

CONDITIONS: Pain
Keywords: Misoprostol; IUD insertion; Nulliparous Women; Contraception; Family Planning; IUD insertion in nulliparous women
MeSH Terms: conditions — Pain | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Experimental): Misoprostol 400 micrograms inserted buccally or vaginally, per the participants desire.
  Interventions: Drug: Misoprostol
- Placebo (Placebo Comparator): Pills which are identical to the study drug in appearance, taste, and smell.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — 400 micrograms inserted buccally or vaginally, per the participants desire prior to the IUD insertion.
  Arms: Misoprostol
Drug: Placebo — Pills which are identical to the study drug in appearance, taste, and smell.
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if using misoprostol makes the intrauterine device insertion easier and less painful in women who have never had a baby.

DETAILED DESCRIPTION:
The Intrauterine Device (IUD) is an excellent contraceptive option because of its ease of use, long term duration (5-10 years), low side-effect profile, and the immediate return to fertility after IUD removal. Despite advantages associated with the IUD, the smaller cervical diameter of nulliparous patients may lead to a more difficult and uncomfortable insertion. Some providers have started pre-medicating nulliparous patients with misoprostol prior to IUD insertion because of the drug's known effect as a cervical ripening agent. Limited evidence is available addressing the effect of misoprostol on patient comfort and provider ease of IUD insertion in nulliparous women. The goal of this study is to evaluate whether using misoprostol as a cervical ripening agent in nulliparous patients eases IUD insertion and decreases pain.

ELIGIBILITY:
Inclusion Criteria:

* 14 years old or older
* Negative pregnancy test
* No prior pregnancies lasting beyond 19 6/7 weeks
* Minimum 2 weeks after spontaneous or medical abortion
* Minimum 4 weeks post 2nd trimester or surgical abortion
* No previous IUD insertions
* No PID in last 3 months
* No current cervicitis
* Willing to follow-up in 1-2 months for an IUD string check

Exclusion Criteria:

* Active cervical infection
* Current pregnancy
* Prior pregnancy beyond 19 6/7 weeks gestation
* Known uterine anomaly
* Fibroid uterus distorting uterine cavity
* Copper allergy/Wilson's Disease (for Paragard)
* Undiagnosed abnormal uterine bleeding
* Cervical or uterine cancer

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 85 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eve Espey, MD/MPH, Principal Investigator — University of New Mexico Department of Obstetrics and Gynecology

REFERENCES:
- [Derived] Turok DK, Espey E, Edelman AB, Lotke PS, Lathrop EH, Teal SB, Jacobson JC, Simonsen SE, Schulz KF. The methodology for developing a prospective meta-analysis in the family planning community. Trials. 2011 Apr 29;12:104. doi: 10.1186/1745-6215-12-104. PMID 21527040

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study design is double-blind randomized controlled trial in which nulliparous women requesting an IUD were randomized to 400 mcg of buccal misoprostol or placebo 2-8 hours before insertion.
Pre-assignment Details: 3 of the 85 enrolled participants were deemed ineligible and not randomized to misoprostol or the placebo group.
Period: IUD Insertion
Arm/Group | Misoprostol | Placebo
Started | 42 | 40
Completed | 40 | 40
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Period: 1-2 Week IUD Check up
Arm/Group | Misoprostol | Placebo
Started | 40 | 40
Completed | 38 | 38
Not Completed | 2 | 2
Not completed — IUD expulsion/removal | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Not Randomized: Women not eligible to continue to randomization.
- Total: Total of all reporting groups
Arm/Group | Misoprostol | Placebo | Not Randomized | Total
Number analyzed (Participants) | 42 | 40 | 3 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.1 (4.3) | 24.1 (4.6) | NA (NA) — Patient data not collected, deemed ineligible after recruitment. | 24.1 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 40 | 3 | 85
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 40 | 3 | 85

OUTCOME MEASURES:

1. Secondary Outcome: Provider Perceived Ease of Insertion on a 100-point Visual Analogue Scale.
Description: Perceived ease of IUD insertion registered on a visual analogue scale (0 = easy, 100 = extremely difficult).
Time Frame: Immediately post IUD insertion
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 40 | 40
units on a scale | 2.2 (2.2) | 2.5 (2.2)

2. Primary Outcome: Patient Perceived Pain on a 100-point Visual Analogue Scale.
Description: Perceived pain was registered on a 100-point visual analogue scale (0 = no pain, 100 = worst pain imaginable) at three time points: prior to IUD insertion, immediately after insertion, and prior to clinic discharge.
Time Frame: Prior to insertion, immediately after insertion, and prior to clinic discharge.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 40 | 40
units on a scale
  Pain perceived prior to insertion | 0.5 (1.2) | 0.8 (1.7)
  Pain perceived immediately after insertion | 5.8 (2.0) | 5.9 (2.0)
  Pain perceived prior to clinic discharge | 3.2 (2.2) | 3.8 (2.7)

ADVERSE EVENTS:
Arm/Group | Misoprostol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No